CLINICAL TRIAL: NCT04649632
Title: Relation Between Dose and Time to Reinjection of Botulinum Toxin-A in Patient With Poststroke Spasticity From a Real-world Healthcare Insurance Database.
Acronym: Relax
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: CLIN-52120-450
Record Dates: First submitted 2020-11-12; First posted 2020-12-02 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Post Stroke Spasticity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No

SUMMARY:
Determining the mean/median time between botulinum toxin-A injection within the treatment of patients with spasticity after stroke in relation to the botulinum toxin dose from a healthcare insurance database in the Netherlands.

ELIGIBILITY:
Inclusion Criteria:

* A patient will be included if he has a diagnosis stroke within the rehabilitation setting and has received at least two injections of botulinum toxin-A: Dysport or Botox

Exclusion Criteria:

* A patient will be excluded if he has been only treated with Xeomin

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients selected from the database claimed within the code 313 will be included in the descriptive analyses.
Sampling Method: Non-Probability Sample
Enrollment: 451 (Actual)
Dates: Start 2020-04-29 (Actual); Primary Completion 2020-09-18 (Actual); Study Completion 2020-09-18 (Actual)

PRIMARY OUTCOMES:
Mean time to next injection per brand | From baseline up to end of data collection (January 2012 up to December 2016)
Median time to next injection per brand | From baseline up to end of data collection (January 2012 up to December 2016)
Dosing of botulinum toxin-A in daily practice in relation to time to next injection | From baseline up to end of data collection (January 2012 up to December 2016)

SECONDARY OUTCOMES:
Average cost per year per brand per patient | From baseline up to end of data collection (January 2012 up to December 2016)
Exploring factors like age, gender, time since diagnosis stroke that influence dosing and time between botulinum toxin-A treatments | From baseline up to end of data collection (January 2012 up to December 2016)
Time interval between 2 injections of the same brand | From baseline up to end of data collection (January 2012 up to December 2016)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (1):
- Ipsen Facility, Hoofddorp, Netherlands